CLINICAL TRIAL: NCT03901391
Title: Prospective Open Label Clinical and Genetic Testing of Patients With Retinitis Pigment
Brief Title: Prospective Open Clinical and Genetic Study of Patients With Retinitis Pigmentosa
Acronym: RU-RP
Status: Completed | Type: Observational
Sponsor: Sensor Technology for Deafblind (Industry)
Collaborators: Central Clinical Hospital under President Affairs (Unknown); Deaf-Blind Support Foundation Con-nection (Unknown); Federal State Budgetary Institution Moscow Helmholtz Eye Research Institute (Unknown); Federal State Budgetary Institution Research Center for Medical Genetics (Unknown); Oftalmic LLC (Unknown); Center for Genetics and Reproductive Medicine Genetico (Unknown)
Responsible Party: Sponsor
Other Study IDs: RU-RP-03-2019
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Retinitis Pigmentosa; Usher Syndromes
MeSH Terms: conditions — Retinitis Pigmentosa; Usher Syndromes | interventions — Exome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retinitis Pigmentosa
  Interventions: Diagnostic Test: Whole Exome Sequencing

INTERVENTIONS:
Diagnostic Test: Whole Exome Sequencing — Whole Exome Sequencing

SUMMARY:
This study is aimed to characterize Russian population of Retinitis Pigmentosa

DETAILED DESCRIPTION:
This study is aimed to characterize Russian population of Retinitis Pigmentosa.

Tasks:

Stage 1. Formation of the primary cohort of patients. Patients pre-recruiting will be performed based on Deaf-Blind Support Foundation "Con-nection" patient database analysis and from references. Patients with clinically confirmed Retinitis pigmentosa will be evaluated according to available data of the clinical examination.

Stage 2. Genetic study of patients. All enrolled patients will undergo single 4 ml peripheral venous blood sampling. DNA will be extracted from leucocytes. DNA samples will be analyzed and placed for long-term storage in liquid nitrogen. Stage 3. Clinical examination of patients.

Each patient will undergo the following diagnostic procedures according to the unified protocol:

* Visometry (with correction and without correction)
* Ophthalmoscopy
* Perimetry
* Optical coherence tomography
* Electroretinography
* Visually evoked potentials
* Refractometry
* Pneumotonometry
* Biomicroscopy
* Any additional examinations and consultations if necessary Medical record will be developed and maintained for each patient consisting results of extended clinical examination.

Statistical and bioinformatic analysis of detected genetic mutations in the study cohort will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patient fulfill the clinical characteristics for Retinitis Pigmentosa (AD, AR, X-linked, sporadic) as defined by the Retinitis pigmentosa consortium
* Results of perimetry for each eye show narrowing for 15 degrees or more.
* Patient is familiar with Participant information sheet
* Patient signed informed consent form

Non-inclusion Criteria:

* Participation in other clinical trials (or administration of investigational drugs) during 3 months prior inclusion
* Any conditions limiting compliance (dementia, neuropsychiatric disease, drug and alcohol abuse etc.)
* Medical history of traumatic injury of eyes, barotrauma, concussion, craniocerebral trauma, cerebrovascular accident
* Congenital multiple development orbit and eye malformations

Exclusion Criteria:

* Patient's refusal from the further participation in the trial
* Decompensated diabetes mellitus
* Severe coronary artery disease
* Chronic infectious disease
* Patients with malignant tumors including postoperative period, patients receiving chemotherapy and/or radiotherapy

Ages: 6 Years to 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: It is assumed that at least 130 patients of the Russian population of men and women aged 6 to 65 years, with verified diagnosis of Retinitis pigmentosa (AD, AR, X-linked or sporadic as defined by the Retinitis pigmentosa consortium), will take part in this research study.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2020-10-19 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
Changes in visual acuity | Up to 4 weeks
  Measured by visual acuity test
Changes in structures of fundus of the eye-1 | Up to 4 weeks
  Measured by ophthalmoscopy
Changes in structures of fundus of the eye-2 | Up to 4 weeks
  Measured by ophthalmoscopy
Changes in visual field | Up to 4 weeks
  Measured by perimetry
Changes in brain visual cortex neural pathways | Up to 4 weeks
  Measured by visually evoked potentials
Changes in electroretinogram | Up to 4 weeks
  Measured by electroretinography
Changes in optical refraction | Up to 4 weeks
  Measured by refractometry
Changes in intraocular pressure | Up to 4 weeks
  Measured by pneumotonometry
Changes in the lens, cornea, anterior segment of the eye | Up to 4 weeks
  Measured by biomicroscopy
Changes in central retinal profile | Up to 4 weeks
  Measured by optical coherent tomography

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry S. Atarshchikov, MD, PhD, Principal Investigator — Central Clinical Hospital under President Affairs
Locations (2):
- Russia (2):
  - Federal State Budgetary Institution "Moscow Helmholtz Research Institute of Eye Diseases" of the Ministry of Health, Moscow
  - Central Clinical Hospital under President Affairs, Moscow

IPD SHARING:
Plan to Share IPD: No